CLINICAL TRIAL: NCT01754792
Title: A Randomized, Double-blind, Placebo-controlled Study on the Influence of Pinitol on Carbohydrate, Lipid and Inflammatory Parameters, Endothelial Function and Oxidative Stress in Diabetic, Impaired and Normal Fasting Glucose Subjects
Brief Title: Effects of Pinitol on Hidrocarbonated Metabolism Parameters in Diabetic, Impaired and Normal Fasting Glucose Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Antonio Hernández Mijares, PhD, MD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WIL-PIN-2012-02
Record Dates: First submitted 2012-12-13; First posted 2012-12-21 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes; Impaired Glucose Tolerance; Healthy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — pinitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal fasting glucose subjects (Experimental): Before pinitol/placebo administration a four weeks run-in period of a healthy diet will be follow for all subjects. After this adaptation period, each subject will be randomized (1:1) into one of two groups: one that received the pinitol-enriched beverage (4 g/day) (n=20), and the other a placebo beverage (n=20) for 12 weeks.
  Interventions: Dietary Supplement: Pinitol
- Impaired fasting glucose subjects (Experimental): Before pinitol/placebo administration a four weeks run-in period of a healthy diet will be follow for all subjects. After this adaptation period, each subject will be randomized (1:1) into one of two groups: one that received the pinitol-enriched beverage (4 g/day) (n=20), and the other a placebo beverage (n=20) for 12 weeks.
  Interventions: Dietary Supplement: Pinitol
- Diabetic subjects (Experimental): Before pinitol/placebo administration a four weeks run-in period of a healthy diet will be follow for all subjects. After this adaptation period, each subject will be randomized (1:1) into one of two groups: one that received the pinitol-enriched beverage (4 g/day) (n=20), and the other a placebo beverage (n=20) for 12 weeks.
  Interventions: Dietary Supplement: Pinitol

INTERVENTIONS:
Dietary Supplement: Pinitol — Fruit Up® (diluted with mineral water to a final volume of 250 ml) will be evaluated, and will be equivalent to an intake of 2 g of pinitol. The placebo beverage will contain equal amounts of non-polyol carbohydrates with similar macronutrient composition and energy intake as that those obtained through the pinitol beverage, but excluding pinitol.
  Other Names: 3-O-methyl-D-chiro-inositol

SUMMARY:
The purpose of this study was to assess whether pinitol improves hidrocarbonated metabolism parameters, and evaluate its effect on oxidative stress and endothelial function in diabetic, impaired and normal fasting glucose subjects.

This was a 3-month randomised, controlled-placebo, parallel trial with a three-arm design. Patients were divided into three groups: diabetic (n=40), impaired fasting glucose (n=40) or normal fasting glucose subjects (n=40), receiving 4 g/day of pinitol/placebo.

ELIGIBILITY:
Inclusion criteria:

* Age range of 18-70 years.
* Normal fasting glucose subjects were diagnosed as fasting glucose <100 mg/dl and HbA1c <5.7%.
* Impaired fasting glucose subjects were diagnosed as fasting glucose between 100 and 125 mg/dl and/or HbA1c between 5.7 and 6.4%.
* Type 2 Diabetes subjects were diagnosed as basal plasma glucose ≥ 126 mg/dl, at least twice, or glucose levels 2 hours after 75 g oral glucose overload ≥ 200 mg/dl (American Diabetes Association)

Exclusion criteria:

* Morbid obesity
* Type 1 diabetes
* Heart, liver, thyroid or kidney untreated disease
* Neoplasic disease
* Hypertriglyceridemia (Triglycerides >400 mg/dl),
* Use of drugs that can influence the inflammatory state or insulin sensitivity (NSAIDs, corticosteroids, antiTNFα) and
* Uncontrolled type 2 diabetes (HbA1c ≥ 8%) or with insulin or intestinal disaccharidase inhibitors (acarbose, miglyol,...) treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To assess hidrocarbonated metabolism parameters before and after pinitol/placebo administration | 3 months
  Blood samples were collected in vacutainer serum separator tubes, after 12- hour overnight fasting, to analyze glucose and insulin concentration at baseline (after a four weeks run-in period of a healthy diet), 6 and 12 weeks after pinitol/placebo administration. Glucose concentrations were measured by means of enzymatic assay in an autoanalyzer. Insulin concentrations were determined by enzyme-linked immunosorbent assay.
  In a representative group of patients of all groups at time 0 and 10 weeks, a 24 hours glucose levels control were assessed (by means of a continuous glucose monitoring system) for 3 days.
  Insulin resistance was estimated by the homeostasis model assessment of insulin resistance (HOMA-IR) index (fasting insulin (μIU/ml) x fasting glucose (mg/dl) /405). Glycosylated hemoglobin (HbA1c) was measured at baseline and 12 weeks in diabetic and impaired fasting glucose subjects.

SECONDARY OUTCOMES:
To evaluate lipid parameters before and after pinitol/placebo administration | 3 months
  Total cholesterol and triglycerides were measured by means of enzymatic assays and HDL cholesterol concentrations were recorded using a direct method with an autoanalyzer. LDL cholesterol concentration was calculated using the Friedewald method. Non-HDL cholesterol concentration was obtained by calculating the difference between total and HDL cholesterol. Atherogenic index of plasma was obtained by calculating the logarithm of the ratio of plasma concentration of triglycerides to HDL-cholesterol. Apolipoprotein A-I and B were determined by immunonephelometry. These parameters were measured at baseline, 6 and 12 weeks after pinitol/placebo administration.
To evaluate inflammatory parameters before and after pinitol/placebo administration | 3 months
  The evaluation of the inflammatory state was assessed by determination of the concentrations of high sensitive C-reactive protein (hsCRP)(by a latexenhanced immunonephelometric assay) and interleukin-6 (IL-6) and tumor necrosis factor alpha (TNF-α) by xMAP Multiplex technology on the Luminex. These parameters were measured at baseline, 6 and 12 weeks after pinitol/placebo administration.
To evaluate endothelial function before and after pinitol/placebo administration | 3 months
  E-selectin, ICAM-1 and VCAM-1 were measured by xMAP Multiplex technology on the Luminex at baseline, 6 and 12 weeks after pinitol/placebo administration
To evaluate oxidative stress on mitochondrial function before and after pinitol/placebo administration | 3 months
  Mitochondrial production of reactive oxygen species, levels of calcium, mitochondrial membrane potential and mitochondrial activity were measured at baseline, 6 and 12 weeks after pinitol/placebo administration

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hernandez, MD, Phd, Principal Investigator — Universtiy of Valencia
Locations (1):
- University Hospital Dr Peset, Valencia, Spain